CLINICAL TRIAL: NCT00163683
Title: The Effect of a Mediterranean Style Diet Versus a Conventional High Carbohydrate, Low Fat Diet on Glycaemic and Lipid Control and on Vascular Inflammatory Markers in People With Newly Diagnosed Type 2 Diabetes
Brief Title: Effects of a Mediterranean Style Diet on Vascular Health in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: A33420
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2005-09

CONDITIONS: Type 2 Diabetes; Coronary Heart Disease
Keywords: Dietary Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Disease | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Dietary Therapy

SUMMARY:
In this study we will compare the effects of a Mediterranean diet, high in fruit and vegetables with the more conventional diet recommended for diabetes therapy (a high carbohydrate, low fat diet) on glycaemic and lipid control and on markers of inflammation, in people with newly diagnosed Type 2 diabetes. The hypothesis is that, over a six-month intervention period, a HVM diet will be more effective than a conventional HCLF diet in improving glycaemic and lipid control, and in reducing markers of vascular inflammation in people with Type 2 diabetes.

DETAILED DESCRIPTION:
Chronic inflammation affecting both small and large blood vessels is an important factor increasing the risk of heart disease in people with Type 2 diabetes. Good markers present in the blood are now available to detect this inflammatory state. Recent evidence suggests that a Mediterranean-type diet, high in plant foods and with monounsaturated fat from olive oil has beneficial effects on blood vessels as well as on blood glucose and blood lipid control.

In this study we will compare the effects of a Mediterranean diet, high in fruit and vegetables with the more conventional diet recommended for diabetes therapy (a high carbohydrate, low fat diet). Twenty-four people with Type 2 diabetes will be randomised to one of these diets and followed for six months. At the end of this time, the effect of the diets on markers for inflammation will be compared.

ELIGIBILITY:
Inclusion Criteria:

-English speaking people with newly diagnosed Type 2 diabetes (within 3-12 months of diagnosis) who are attending the Alfred Hospital, Diabetes Education Outpatient Clinic.

Exclusion Criteria:

* age <30 years or > 75 years;
* body mass index (BMI) < 25 kg/m2 or >37 kg/m2;
* on corticosteroid or insulin therapy;
* presence of established renal and/or liver disease (serum creatinine more than 0.12 mmol/L/albumin excretion rate greater than 300 µg per minute or ALT more than twice the upper limit of normal respectively).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The primary outcomes include: HBAIc and lipids (Cholesterol, HDL-cholesterol, Triglycerides) at study entry and 6 months after dietary intervention

SECONDARY OUTCOMES:
Key secondary outcomes include: TNF-a, IL-6, High sensitivity CRP, plasma carotenoids and serum fatty acids.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel M Stoney, PhD, Principal Investigator — Alfred Hospital, Melbourne, AUSTRALIA; Karen Z Walker, PhD, Study Director — Monash University; Duncan Topliss, FRACP, Study Director — Alfred Hospital, Melbourne, AUSTRALIA
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia